CLINICAL TRIAL: NCT01055470
Title: Open, Randomized, Controlled Clinical Trial of Lornoxicam as Compared to Diclofenac in Osteoarthritis of Knee Joint in Patients of Tertiary Care Hospital of Gujarat.
Brief Title: Comparative Clinical Trial of Lornoxicam to Diclofenac in Patients of Osteoarthritis of Knee Joint.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Bhavnagar (Other)
Responsible Party: Dr. C. B. Tripathi, Professor and Head , Department of Pharmacology, Government Medical College, Bhavnagar-364001, Gujarat, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pharmacol no.02 /2008 Research
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2010-01

CONDITIONS: Osteoarthritis of Knee Joint
MeSH Terms: interventions — Diclofenac; lornoxicam

ARMS (2):
- Diclofenac (Active Comparator): Tab.Diclofenac 50 mg ,Orally, 12 hrly in morning and in evening after taking food for 3 months.
  Interventions: Drug: Diclofenac
- Lornoxicam (Experimental): Tab. Lornoxicam 4 mg , orally, 8 hourly after taking food in morning , in noon and evening for 3 months.
  Interventions: Drug: Lornoxicam

INTERVENTIONS:
Drug: Diclofenac — Tab. Diclofenac 50 mg 12 hrly, orally, in morning and in evening after taking food for 3 months.
  Arms: Diclofenac
Drug: Lornoxicam — Tab. Lornoxicam 4 mg , orally, 8 hourly after taking food in morning , in noon and evening for 3 months.
  Arms: Lornoxicam

SUMMARY:
The purpose of this study was to compare the pain relieving action of the lornoxicam and diclofenac in patients of OA knee.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patient aged between 25 to 65 yrs of either gender suffering from osteoarthritis of knee according to criteria given by American College of Rheumatology
* Informed consent obtained from the patient.

Exclusion Criteria:

* Patients with any other systemic llness,
* Patients with pregnancy and lactation,
* Patients taking other drugs like lithium[4], digoxin, methotrexate, anticoagulants, antidiabetics, diuretics,
* Patients with H/O hypersensitivity to NSAIDs,
* Patients who had consumed any analgesics in last 1 month

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Difference in reduction in reading of Wong Baker face pain scale and in time of 100 meters walking test | 3 months

SECONDARY OUTCOMES:
To monitor side effects of study drugs. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Vishalkumar Kishorbhai Vadgama, M.B;B.S., Principal Investigator — Department of Pharmacology, Government Medical College, Bhavnagar-364001, Gujarat, India; Dr. Chandrabhanu Rajkishore Tripathi, M.D. (Pharmacology), Study Chair — Proffessor and Head, Department of Pharmacology, Government Medical College, Bhavnagar-364001, Gujarat, India
Locations (1):
- Sir Takthasinhji General Hospital, Bhavnagar, Gujarat, India